CLINICAL TRIAL: NCT02486432
Title: A Single Period Investigation to Assess the Tolerability of Healthy Subjects to Oral Sinemet® (Levodopa/Carbidopa) Doses Administered Using a Divided Dose Approach
Brief Title: A Single Period Investigation to Assess the Tolerability of Healthy Subjects to Oral Sinemet® (Levodopa/Carbidopa)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ND0612-013
Record Dates: First submitted 2015-06-22; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm Levodopa/Carbidopa (Experimental): The intervention is dosing with Sinemet® which is an oral tablet containing Levodopa/Carbidopa. Oral administration of 2 × 12.5 mg/50 mg Sinemet® tablet containing 13.5 mg carbidopa (equivalent to 12.5 mg anhydrous carbidopa) and 50 mg levodopa three times a day on Day -1 with 240 mL water Oral administration of 1 × 12.5 mg/50 mg Sinemet® tablets containing 13.5 mg carbidopa (equivalent to 12.5 mg of anhydrous carbidopa) and 50 mg levodopa administered with 100 mL water every hour for 16 hours on Day 1
  Interventions: Drug: Levodopa/Carbidopa (Sinemet)

INTERVENTIONS:
Drug: Levodopa/Carbidopa (Sinemet) — Oral administration of 2 × 12.5 mg/50 mg Sinemet® tablet containing 13.5 mg carbidopa (equivalent to 12.5 mg anhydrous carbidopa) and 50 mg levodopa three times a day on Day -1 with 240 mL water Oral administration of 1 × 12.5 mg/50 mg Sinemet® tablets containing 13.5 mg carbidopa (equivalent to 12.5 mg of anhydrous carbidopa) and 50 mg levodopa administered with 100 mL water every hour for 16 hours on Day 1
  Other Names: Sinemet

SUMMARY:
A Single Period Investigation to Assess the Tolerability of Healthy Subjects to Oral Sinemet® (Levodopa/Carbidopa) Doses Administered Using a Divided Dose Approach

DETAILED DESCRIPTION:
This is a single centre, open-label, single period study in healthy subjects. Each subject will receive the following regimen:

On Day -2, 10 mg domperidone administered every 8 hours 3 times a day (for illustrative purposes, dosing at 07:30, 15:30 and 23:30) On Day -1, 3 doses of 100 mg Sinemet® (every 8 hours) administered as 2 × Sinemet® 12.5 mg/50 mg tablets containing 13.5 mg carbidopa (equivalent to 12.5 mg anhydrous carbidopa) and 50 mg levodopa. Subjects will receive concomitant 10 mg domperidone 30 minutes before every Sinemet® dose.

On Day 1, Sinemet® 12.5 mg/50 mg containing 13.5 mg carbidopa (equivalent to 12.5 mg of anhydrous carbidopa) and 50 mg levodopa administered every hour for 16 consecutive doses (total dose of 800 mg). Subjects will also receive concomitant domperidone up to 20 mg 30 minutes before the first Sinemet® 50 mg dose and every 8 hours (total of 3 doses) after treatment initiation.

It is planned to enrol 6 subjects to ensure there are 6 evaluable subjects. A subject is considered to be evaluable if they have received all 16 Sinemet® 50 mg doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Age 40 to 65 years of age
3. Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
7. Females of childbearing potential who are pregnant or lactating (female subjects must have a negative urine pregnancy test at admission)
8. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1)
9. Positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1)
10. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
11. History of cardiovascular, renal, hepatic, chronic respiratory or GI disease as judged by the investigator
12. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
13. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
14. Donation or loss of greater than 400 mL of blood within the previous 3 months
15. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol, hormone replacement therapy and hormonal contraception) or herbal remedies in the 14 days before IMP administration (See Section 11.4)
16. Use of any non-selective monoamine oxidase (MAO) inhibitors within 2 weeks of screening
17. History or presence of glaucoma
18. History or presence of suspicious undiagnosed skin lesions or a history of melanoma
19. Any history of psychoses or seizure
20. Known hypersensitivity to Sinemet® or domperidone or any of the excipients
21. Any history or presence of Prolactin-releasing pituitary tumour (prolactinoma)
22. Any medical history of GI haemorrhage, mechanical obstruction or perforation
23. Any history of moderate or severe hepatic impairment
24. Subjects with clinically significant liver function tests
25. Subjects with QTc > 450 ms at screening Sponsor/Quotient Clinical Confidential Protocol ND0612-013 (QCL117546) Version 1.0 02 FEB 2015 Page 23 of 42
26. Subjects with significant electrolyte disturbances
27. Subjects with any underlying cardiac disease
28. Subjects who have received QT-prolonging drugs or potent cytochrome P450 (CYP) 3A4 inhibitors within 4 weeks of screening
29. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The objective of the study is to provide safety and tolerability information for oral doses of levodopa and carbidopa administered as a divided dose. | 5 weeks
  Safety and tolerability will be assessed by: adverse events (AEs), physical examination, safety laboratory tests, vital signs and electrocardiograms (ECGs).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, MRCS, Principal Investigator — Quotient Clinical Mere Way Ruddington Fields Ruddington Nottingham NG11 6JS, UK